CLINICAL TRIAL: NCT00514202
Title: Dextroamphetamine Treatment for Comorbid Cocaine Dependence and ADHD
Brief Title: Pilot Study Examining Effect for Dextroamphetamine to Treat Cocaine Dependence Plus Attention-deficit Hyperactivity Disorder (ADHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left UTHSC-Houston
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-07-0024; P50DA009262 (NIH)
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Cocaine-Related Disorders; Substance-Related Disorders
Keywords: cocaine; ADHD; attention; hyperactivity; drug; dependence
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Cocaine-Related Disorders; Substance-Related Disorders; Spasm | interventions — Amphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo plus cognitive behavioral therapy
  Interventions: Drug: Placebo
- 2 (Experimental): Dextroamphetamine SR (60 mg/kg) plus cognitive behavioral therapy
  Interventions: Drug: Dextroamphetamine SR

INTERVENTIONS:
Drug: Placebo — matched placebo
  Arms: 1
Drug: Dextroamphetamine SR — 60 mg/day
  Other Names: Dexedrine Spansules
  Arms: 2

SUMMARY:
Dextroamphetamine is commonly used to treat ADHD, and recent evidence suggests that this medication may decrease drug use in individuals dependent on cocaine. Thus, the present pilot study will determine the ability of dextroamphetamine to treat individuals with both cocaine dependence and ADHD.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled pilot study will determine the ability of dextroamphetamine to treat comorbid cocaine dependence and ADHD. Participants will be randomly assigned on receive placebo or Dextroamphetamine SR (60 mg/day) during a 12-week study period. All participants will receive weekly cognitive behavioral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Generally good health except for problems related to drug use
* Meet DSM criteria for cocaine dependence and ADHD
* Have stable living situation

Exclusion Criteria:

* DSM diagnosis for current psychotic, anxiety disorders as well as current substance dependence (with the exception of marijuana and nicotine)
* Current use of prescription medications
* Females who are currently pregnant or nursing
* History of significant acute or chronic physical illness
* History of or current liver disease
* Existing cardiovascular disease
* Plans to leave metropolitan area within 3 months
* Probation or parole with constraints that preclude full study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Substance use | Duration of study
ADHD symptoms | Duration of study

SECONDARY OUTCOMES:
Treatment retention | Duration of study
Cocaine craving | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: David V Herin, Ph.D, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States